CLINICAL TRIAL: NCT06428903
Title: A Comparison Study of ADC189 Bioavailability Between Tablet and Granule in Healthy Chinese Adult Male Subjects, and the Safety and Pharmacokinetics of Ultra-high Dose ADC189
Brief Title: Comparative Bioavailability Study of Tablet and Granule Formulations of ADC189 and the Study of Ultra-high Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiaxing AnDiCon Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ADC-DNXV-189-GR
Record Dates: First submitted 2024-05-19; First posted 2024-05-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADC189 tablet Group A (Experimental): 16 patients.
  Interventions: Drug: ADC189 tablet; Drug: ADC189 granules
- ADC189 granules Group B (Experimental): 16 patients.
  Interventions: Drug: ADC189 tablet; Drug: ADC189 granules
- ADC189 180mg Group (Experimental): 8 patients.
  Interventions: Drug: ADC189 180mg

INTERVENTIONS:
Drug: ADC189 tablet — ADC189 tablet, 45 mg, single oral dose in each Group. (Part 1 study)
  Arms: ADC189 granules Group B; ADC189 tablet Group A
Drug: ADC189 granules — ADC189 granules, 45 mg, single oral dose in each Group. (Part 1 study)
  Arms: ADC189 granules Group B; ADC189 tablet Group A
Drug: ADC189 180mg — ADC189 tablet, 180 mg, single oral dose. (Part 2 study)
  Arms: ADC189 180mg Group

SUMMARY:
Part 1 of this study will compare the pharmacokinetic performance of tablet and granule formulations of ADC189 under fasted conditions in healthy volunteers. A randomized, two-period, two-treatment crossover design is used. In each period, each volunteer will receive a single oral dose of the tablet or granule formulation without food.

The purpose of Part 2 study is to determine the safety and pharmacokinetics of ultra high dose of ADC189 in healthy subjects.

DETAILED DESCRIPTION:
In Part 1 study, a total of 32 subjects were randomly divided into two groups, A and B, with 16 subjects in each group. After a 28-day screening period, on the first day of Period 1 (D1), subjects in group A took ADC189 granules (a single oral dose, 45mg), and subjects in group B took ADC189 tablets (a single oral dose, 45mg), all subjects were under fasted conditon. In Period 2, two groups will change to the fomulation which is different in Period 1 respectively, and all the steps will keep the same as Period 1. Each period lasts for 15 days, and have a 7-day interval between 2 periods. Blood samples will be taken, pharmacokinetic and saftey profiles will be observed.

In Part 2 study, the ultra high dose of ADC189 (a single oral dose, 180mg) will applied in 8 healty adult male subjects. The pharmacokinetic and saftey profiles will be observed during the following 15 days, and blood sample will be taken.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male subjects aged 18-45 years old
* 2. Male subjects weight over 50 kg

Exclusion Criteria:

* 1. Any other clinically relevant abnormalities, concomitant diseases or ongoing medical conditions
* 2. Have a history of drug abuse in the past five years or use drugs in the three months prior to screening
* 3. Blood donation or blood loss > 400 mL in 3 months before screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
ADC189 Granules | 15 days
  ADC189 plasma exposure, area under the concentration-time curve
ADC189 Tablet | 15 days
  ADC189 plasma exposure, area under the concentration-time curve
ADC189 Ultra high dose | 15 days
  Single dose of 180mg ADC189 tablet plasma exposure, area under the concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Zhao Wei, Jinan, Shang Dong, China

IPD SHARING:
Plan to Share IPD: No